CLINICAL TRIAL: NCT04129697
Title: Intratympanic Dexamethasone or Methylprednisolone for Sudden Hearing Loss as a Salvage Treatment: a Randomized, Double-blind, Multi-center Study
Brief Title: Intratympanic Steroids for Sudden Hearing Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019SHLRCT
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Dexamethasone or Methylprednisolone; Sudden Hearing Loss; Intratympanic Steroid
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone or Methylprednisolone
- Methylprednisolone (Active Comparator)
  Interventions: Drug: Dexamethasone or Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone or Methylprednisolone — steroids

SUMMARY:
For patients with sudden hearing loss, the initial treatment is not usually effective. We use Dexamethasone or Methylprednisolone to be an Intratympanic steroid administration as a salvage treatment. An randomized, double-blind, multi-center study is designed to find the difference between Dexamethasone or Methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

sudden hearing loss and initial treatment is not effective

Exclusion Criteria:

the patients refused intratympanic steroids treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
hearing | six month
  the hearing level after treatment

IPD SHARING:
Plan to Share IPD: Undecided
The results of the study could be shared with other researchers